CLINICAL TRIAL: NCT00154674
Title: Safety and Feasibility of Endovascular Cooling Device in Patients With Hypothermic Cardiopulmonary Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25MD03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2004-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

INTERVENTIONS:
Device: ICY catheter, Thermoguard device

SUMMARY:
Hypothermic resuscitation is proven to be benefit to the cardiac origin cardiac arrest patients for it improve brain recovery dramatically. However, traditional cooling devices and methods, most external cooling methods, include ice blanket, cooling helmet, or ice packing lower the body temperature slowly or inefficiently which make many emergency physicians hesitate to perform hypothermic resuscitation. To improve and promote the practice of hypothermia resuscitation, more efficient temperature control method is necessary. We conduct this clinical trial to evaluate the safety and feasibility of internal cooling catheter and temperature regulatory device, which is approved by FDA in neurologic ICU for temperature control, in the cardiac arrest patients.

DETAILED DESCRIPTION:
We recruited successful resuscitated nontraumatic cardiac arrest adult patients in the emergency department to evaluate the safety and feasibility of application those invasive internal temperature regulator devices. Internal cooling catheter, "ICY" , and thermal regulator device, "Coolguard 2000" are applied to the patients from femoral vein. WE definite 4 stages according to the temperature during the clinical trial: "The Cooling Phase", "Hypothermia phase", "Rewarming phase", and "Postrewarming phase". The temperature is lowed or elevated by the rate 0.5C/hr during the Cooling and Rewarming Phase, and it is maintained 33 +/- 1 C during hypothermia phase for 12 hours according to the comment of ACLS. To understand the safety and feasibility, regular blood sampling, bedside EEG and vital monitors, and special sheets are designed to document the every reasons, time points or every clinical events during hypothermia therapy. The patients is observed until rewarming finish for 48 hours or till death if expired during post-resuscitation hypothermia therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic collapsed patients, whose pulsation continues and persists more than 5 minutes after return of spontaneous circulation from cardiopulmonary resuscitation and consciousness level is less than GCS 5 points.

Exclusion Criteria:

* 1. Age > 78 y/o or < 18 y/o 2. Core temperature< 34℃or > 38 ℃ after resuscitation 3. Pregnancy 4. Underline terminal malignancy disorder or refuse aggressive treatment cancer patient 5. Massive bleeding, known coagulopathy, or received regular anticoagulant medication 6. Persisted hypotension ( mean arterial BP < 60 mmHg) after resuscitation even under inotropic agents 7. No bed available in ICU

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-04; Study Completion 2005-10

PRIMARY OUTCOMES:
complications and feasibility of endovascular cooling device

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jone Chen, PHD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan